CLINICAL TRIAL: NCT05963789
Title: Efficacy of Cervical Proprioceptive Exercises in Treating Shoulder Impingement Syndrome
Brief Title: Cervical Proprioception and Shoulder Impingement Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma eldesoky, Physiotherapist at 23rd of July hospital, PhD candidate physiotherapy, Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004185
Record Dates: First submitted 2023-05-12; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Shoulder Impingement; Shoulder Pain
Keywords: Cervical Proprioceptive Exercises; Shoulder pain; Shoulder disability; Shoulder proprioception
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A or cervical proprioception group CPG (Experimental): Patients will receive traditional exercises for shoulder impingement plus cervical proprioception exercises using laser pointer
  Interventions: Other: Cervical proprioceptive training
- Group B or control group CG (Active Comparator): Patients will receive traditional exercises for shoulder impingement (stretching, strengthening, stabilization)
  Interventions: Other: Traditional exercises

INTERVENTIONS:
Other: Cervical proprioceptive training — Cervical proprioceptive training: The laser pointer will fixed on the highest point of the subject head with a band, patients sit upright on a chair and kept their head at the neutral position, while setting the laser light at the point on the wall in front of them. From this position, patients will be asked to flex, extend and rotate their head and then return to the neutral position. This training commenced with open eyes and then progress with closed eyes, tracing a pattern and standing position.
  Other Names: Traditional exercises
  Arms: Group A or cervical proprioception group CPG
Other: Traditional exercises — Stretching posterior shoulder capsule Strengthening scapular muscles Shoulder stabilization PNF
  Arms: Group B or control group CG

SUMMARY:
The aim of this study will be to investigate the role of cervical proprioceptive training on shoulder proprioception, pain, and disability in shoulder impingement syndrome patients

DETAILED DESCRIPTION:
Study design: This study will be randomized controlled trial 1. Participants: fifty males and females patients with functional shoulder impingement, aged from 25-40 years with BMI <32kg/m2. Sample size calculation: The sample size is 50 patients in the 2 experimental groups based on power analysis done calculating effect size from outcomes of previous study (effect size d of 0.82 for shoulder proprioception) . Power analysis was done using G*power software. Power set to (0.8), significance (0.05). Procedture: First, eligible patients will have the purpose of the study and the procedures fully explained. Then, patients will be asked to participate in the study. If they accepted, an informed consent form will be signed and randomly assigned in one of two groups. Afterwards Prior to starting of the study each patient will sign informed consent Patients will be assigned to two groups randomly (by closed envelope method). All subjects will be evaluated for their shoulder pain, disability level, and proprioception. All patients will be tested before and after the treatment program (12 treatment sessions, 3 sessions per week for 4 weeks) Conventional Physical therapy: a. Cross-body stretch b. Sleeper stretch. c. Prone extension with an externally rotated (thumb out) position d. Prone horizontal abduction e. PNF D2 flexion For intervention group it will take Cervical proprioceptive training Retraining joint position sense will be done with a laser pointer. The laser pointer will fixed on the highest point of the subject head with a band. In this exercise, patients sit upright on a chair and kept their head at the neutral position while setting the laser light at the point on the wall in front of them. From this position, patients will be asked to flex, extend and rotate their head and then return to the neutral position. This training commenced with open eyes and then progress with closed eyes, tracing a pattern and standing position . Temporary reproduction of dizziness is acceptable however exacerbation of neck pain or headache is not acceptable. If this occurs the exercises should be modified by decreasing the number of repetitions or altering the patient position to a more supported position. Progression of exercise set can be achieved by altering the duration, repetitions and the degree of difficulty of the task. Exercises can also be progressed by performing activities such as an eye task or cervical JPS practice while sitting on an unstable surface or while standing with the feet in an unstable base of support for example, heel toe stance, or while walking .

ELIGIBILITY:
Inclusion Criteria:

* Shoulder impingement syndrome (defined as patients with at least 3 out of the following 6 criteria; Positive "Neer's sign", Positive "Hawkins' sign", Pain with active shoulder elevation in the scapular plane, Pain in the C5-C6 dermatome, Pain with palpation of the rotator cuff tendons, and Pain with resisted isometric abduction.
* Patients with positive apprehension sign for anterior instability.
* Age 25-40years. 4-BMI<32 kg/m2.

Exclusion Criteria:

* Shoulder osteoarthritis

  * Shoulder trauma
* Shoulder infection
* Intra-articular corticosteroid or hyaluronic acid injection within the last 3 months.
* Previous surgery of the affected shoulder. - Symptomatic cervical pathology.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Shoulder proprioception | 4 weeks
  Joint position sense (Active joint angular reproduction) will be measured with bubble inclinometer during shoulder IR and ER 300 as reference angles from modified neutral position of the arm (shoulder abducted 30O, horizontally adducted 30O and elbow flexed 90o), visual cues are often negated.

SECONDARY OUTCOMES:
Pain and disability | 4 weeks
  Participants will fill the questionnaire of shoulder pain and disability index (SPADI, . Scores will be calculated as follow, scores in all questions will be added in each section separately.
Cervical proprioception | 4 weeks
  Cervical active JPS will be measured using Revel's laser method to record joint position error (JPE). Cervical Joint Position Error (JPE) is the ability to relocate the head to a beginning position following a dynamic active cervical range of motion.

CONTACTS AND LOCATIONS:
Overall Officials: Abdel Majeed, Principal Investigator — Professor at orthopedic department, faculty of physical therapy, Cairo University
Locations (1):
- Fatma eldesoky Ramadan, Cairo, Cairo Governorate, Egypt